CLINICAL TRIAL: NCT04860401
Title: A Miniaturized Device to Non-invasively Measure the Oxygenation and Hemoglobin Concentration in the Brain Using Near-infrared Spectroscopy
Brief Title: OxyPrem Validation Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The substudy in premature infants was completed. The substudy in adult volunteers will not be continued, due to previous delays.
Sponsor: Hans Ulrich Bucher (Other)
Responsible Party: Sponsor-Investigator, Hans Ulrich Bucher, Principal Investigator, University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PB_2016-00395
Record Dates: First submitted 2021-04-15; First posted 2021-04-27 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Tissue Oxygenation Measurement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- precision and accuracy study (Experimental): precision and accuracy of Oxyprem are studied
  Interventions: Device: Measurement of tissue oxygenation with novel diagnostic near-infrared spectroscopy device (OxyPrem) (no clinical decisions based on oxygenation levels)

INTERVENTIONS:
Device: Measurement of tissue oxygenation with novel diagnostic near-infrared spectroscopy device (OxyPrem) (no clinical decisions based on oxygenation levels) — The precision of OxyPrem is assessed by repeated measurements of tissue oxygenation and hemoglobin concentration. The accuracy of OxyPrem is assessed by comparing the measurement data to those acquired simultaneously by established NIRS devices and standard clinical monitoring devices. In substudy 1, healthy adult subjects are enrolled, in substudy 2, measurements are conducted on preterm neonates.

SUMMARY:
The precision of the novel diagnostic near-infrared spectroscopy (NIRS) device for the measurement of tissue oxygenation and hemoglobin concentration (OxyPrem) is assessed by repeated measurements. The accuracy of OxyPrem is assessed by comparing the measurement data to those acquired simultaneously by established NIRS devices and standard clinical monitoring devices. In substudy 1, healthy adult subjects are enrolled, in substudy 2, measurements are conducted on preterm neonates.

ELIGIBILITY:
Substudy 1 (healthy adult volunteers)

Inclusion Criteria:

* Healthy adult
* Signed informed consent

Exclusion Criteria:

* Dense black hair at the location of measurement
* Neurological diseases.

Substudy 2 (preterm infants)

Inclusion Criteria:

* Pre-term neonates (gestational age at birth less than 37 weeks)
* Signed informed consent by at least one parent

Exclusion Criteria:

* Clinically instability
* Malformations

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2010-08-04 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-06-21 (Actual)

PRIMARY OUTCOMES:
Standard deviation of repeated StO2 level measurements (precision) | baseline
  The precision of the StO2 measurement is the reproducibility within multiple consecutive measurements under similar conditions, expressed as the standard deviation of repeated measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Bucher, Prof.em., Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland